CLINICAL TRIAL: NCT05498597
Title: First-in-Human, Phase 1 Study of AMT-151, an Anti-Folate Receptor Alpha Antibody-Drug Conjugate, in Patients With Selected Advanced Solid Tumours
Brief Title: AMT-151 in Patients With Selected Advanced Solid Tumours
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Multitude Therapeutics Inc. (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMT-151-01
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor; Advanced Cancer; Advanced Carcinoma; Ovarian Cancer; Ovarian Carcinoma; Ovarian Epithelial Cancer; Ovarian Endometrioid Adenocarcinoma; Endometrial Cancer; Endometrial Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Endometrioid Adenocarcinoma; Endometrial Clear Cell Adenocarcinoma; Lung Adenocarcinoma; Triple Negative Breast Cancer; Pancreatic Ductal Adenocarcinoma; Malignant Pleural Mesothelioma; Ovarian Clear Cell Carcinoma; Ovarian Clear Cell Adenocarcinoma; Ovarian Mucinous Adenocarcinoma
Keywords: Carcinoma; Cancer; Antibody-Drug Conjugate; Folate Receptor Alpha
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Endometrial Neoplasms; Adenocarcinoma of Lung; Triple Negative Breast Neoplasms; Mesothelioma, Malignant; Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMT-151 Dose Escalation (Experimental)
  Interventions: Drug: AMT-151

INTERVENTIONS:
Drug: AMT-151 — Administered intravenously

SUMMARY:
This first-in-human study will evaluate the Maximum Tolerated Dose (MTD) / the Recommended Phase 2 Dose (RP2D), safety, tolerability, anti-tumor activity, pharmacokinetics, pharmacodynamics and immunogenicity of AMT-151, a novel antibody-drug conjugate against folate receptor alpha, in patients with selected advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must be willing and able to sign the Informed Consent Form, and to adhere to the study visit schedule and other protocol requirements.
* Age ≥18 years (at the time consent is obtained).
* Patients with the following histologically confirmed, advanced cancer diagnoses:

  1. Serous, endometrioid, clear-cell, or mucinous epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
  2. Serous, endometrioid, or clear-cell endometrial cancer.
  3. Adenocarcinoma of the lung.
  4. Triple-negative breast cancer.
  5. Pancreatic ductal adenocarcinoma.
  6. Malignant pleural mesothelioma.
* Patients who have undergone any number of prior systemic therapies and have radiologically or clinically determined progressive disease during or after their most recent line of therapy, and for whom no further standard therapy is available, or who are intolerable to standard therapy.
* Patients must have at least one measurable or non-measurable lesion as per RECIST version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate function of bone marrow, liver, kidneys, heart.
* Both male and female patients must agree to use effective contraceptive methods.
* Women of child-bearing potential (WCBP) must have a negative serum pregnancy test.
* Availability of tumour tissue sample (either an archival specimen or a fresh biopsy material) at screening.

Key Exclusion Criteria:

* Prior treatment with any agent targeting Folate Receptor Alpha.
* Active central nervous system metastasis.
* Persistent toxicities from previous systemic anti-neoplastic treatments of Grade >1.
* Systemic anti-neoplastic therapy within five half-lives or 21 days, whichever is shorter, prior to the first dose of the study drug.
* Radiotherapy to lung field at a total radiation dose of >= 20 Gy within 6 months, wide-field radiotherapy (>30% of marrow-bearing bones) within 28 days, or focal radiation for analgesic purpose or for lytic lesions at risk of fracture within 14 days prior to the first dose of the study drug, or no recovery from side effects of such intervention.
* Major surgery (not including placement of vascular access device or tumor biopsies) within 28 days prior to the first dose of the study drug, or no recovery from side effects of such intervention.
* Prior allogeneic or autologous bone marrow transplantation.
* Significant cardiac or lung disease, active or chronic ocular disorders, thromboembolic or cerebrovascular events within 6 months prior to the first dose of the study drug, acute and/or clinically significant bacterial, fungal, or viral infection.
* Pregnant or breast-feeding females.

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 24 months
  The RP2D will be determined using dose limiting toxicities (DLTs) and all other available study data
Maximum Tolerated Dose (MTD) | Up to 24 months
  The MTD will be determined using DLTs
Incidence of Adverse Events | Up to 24 months
  Safety and tolerability profile assessed by the Common Terminology Criteria for Adverse Events v5.0

SECONDARY OUTCOMES:
Overall Response Rate (ORR) according to the Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 | Up to 24 months
  Proportion of patients achieving Complete Response (CR) or Partial Response (PR)
Disease Control Rate (DCR) according to the RECIST v1.1 | Up to 24 months
  Proportion of patients achieving CR, PR or Stable Disease (SD)
Progression-free Survival (PFS) | Up to 24 months
  Time from date of start of treatment to date of the first progression or death, whichever occurs first.
Time to Treatment Response (TTR) | Up to 24 months
  Time from date of start of treatment to date of the first assessment of response (PR or CR)
Duration of Response (DoR) | Up to 24 months
  Time from date of first assessment of response (CR or PR) to date of the first progression or death, whichever occurs first
Overall Survival (OS) | Up to 24 months
  Time from date of start of treatment to date of death
Concentration of anti-drug antibodies (ADA) | Up to 24 months
  Immunogenicity profile characterized by concentration of ADAs
Maximum observed concentration (C[max]) | Up to 24 months
  Pharmacokinetic profile characterized by the maximum observed concentration (C[max]) of AMT-151
Area under the curve (AUC) | Up to 24 months
  Pharmacokinetic profile characterized by the area under the curve (AUC) of AMT-151
Terminal half-life (t[1/2]) | Up to 24 months
  Pharmacokinetic profile characterized by the terminal half-life (t[1/2]) of AMT-151
Time to maximum concentration (Tmax) | Up to 24 months
  Pharmacokinetic profile characterized by the time to maximum concentration (Tmax) of AMT-151

CONTACTS AND LOCATIONS:
Overall Officials: Sarwan Bishnoi, Principal Investigator — Cancer Research SA; Richardson Gary, Principal Investigator — Cabrini Malvern Hospital; Steven Kao, Principal Investigator — Chris O'Brien Lifehouse; Catherine Shannon, Principal Investigator — Mater Cancer Care Centre; Jermaine Coward, Principal Investigator — ICON Cancer Centre; Mihitha Ariyapperuma, Principal Investigator — One Clinical Research (OCR)
Locations (9):
- Australia (6):
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - ICON Cancer Centre, Brisbane, Queensland
  - Mater Cancer Care Centre, South Brisbane, Queensland
  - Cancer Research SA, Adelaide, South Australia
  - Cabrini Malvern Hospital, Malvern, Victoria
  - One Clinical Research (OCR), Perth, Western Australia
- China (3):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanghai Tumor Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No